CLINICAL TRIAL: NCT06743152
Title: Comparison of the Effects of Synchronous and Asynchronous Telerehabilitation on Fatigue and Functional Capacity in Juvenile Familial Mediterranean Fever Patients
Brief Title: Comparison of the Effects of Synchronous and Asynchronous Telerehabilitation in Patients with Juvenile Familial Mediterranean Fever
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Namli, MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANamli
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Familial Mediterranean Fever (FMF ); Exercise; Telerehabilitation
MeSH Terms: conditions — Familial Mediterranean Fever; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- synchronous telerehabilitation group (Experimental): Synchronous telerehabilitation group will be applied a synchronous supervised online exercise program under the supervision of a physiotherapist
  Interventions: Behavioral: Synchronous exercise program
- Asynchronous telerehabilitation group (Experimental): Asynchronous telerehabilitation group will be applied an asynchronous video-based exercise program.
  Interventions: Behavioral: Asynchronous exercise group

INTERVENTIONS:
Behavioral: Synchronous exercise program — The synchronous exercise group will be conducted online with synchronous supervision under the supervision of a physiotherapist. The exercise program will be performed for 8 weeks, 2 days a week. In the exercise program, 3 sets, 8 repetitions in 1 set will be progressed to 10-12-15-20-25 repetitions according to tolerance. There will be a 1-2 minute rest between sets.
  Arms: synchronous telerehabilitation group
Behavioral: Asynchronous exercise group — The Asynchronous Exercise Group will be conducted with a video-based structured exercise program. For the asynchronous video-based group, a closed channel will be created on Youtube that only patients can access, and the exercises will be uploaded to the system asynchronously. In the asynchronous exercise group, how each exercise is performed will be shown in detail by the physiotherapist in the video content.
  Arms: Asynchronous telerehabilitation group

SUMMARY:
Our study will be randomized controlled. Familial Mediterranean Fever patients between the ages of 12-18 will be included in the study and will be divided into 2 groups. The first group will be applied a synchronous supervised online exercise program under the supervision of a physiotherapist, and the second group will be applied an asynchronous video-based exercise program. The exercise program will be carried out for 8 weeks, 2 days a week. There will be 3 sets, 8 repetitions in 1 set in the exercise program and will be progressed according to tolerance. In the exercise program, the synchronous group will perform the exercises with the supervision of a physiotherapist via the Zoom application, while the asynchronous video-based group will upload the exercises to the system asynchronously via a channel on YouTube that only patients can access. Feedback will be received from the asynchronous group by phone. Our exercise program will be organized with the progression of exercises such as squat, lunge, stepping, running in place and jumping. The primary outcome measures of the study are the evaluation of fatigue (VAS) and functional capacity (6-Minute Walking Test). Our secondary outcome measures are the evaluation of pain, balance, physical fitness and walking. For the assessment of fatigue: Visual Analog Scale (VAS), PedsQL Multidimensional Fatigue Scale, Fatigue Severity Scale; For the assessment of functional capacity: 6 Minute Walk Test, 30 sec Sit-to-Stand Test, 10-Step Climbing Test, Pacer aebonic fitness test, Half Squat Test; For the assessment of balance: One-Leg Stand Test, Functional Forward Reach Test, Kinvent (K-plate)-K Force measurement evaluation set, Digitsole Smart Insole System for the assessment of walking; For the assessment of physical fitness: FitnessGram test battery; For the assessment of pain: VAS will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12-18
* The parent's willingness to have their child participate in the study
* Being diagnosed with FMF at least 6 months ago
* Being in an attack-free period
* Have an internet access
* Being able to use a computer, tablet or smartphone
* Have access to a technological device with a camera, microphone and speaker output
* Being willing to participate in the study

Exclusion Criteria:

* Having any musculoskeletal disease or orthopedic, neurological, psychological disease that may prevent participation in exercise
* Acute pain for any reason
* Development of amyloidosis

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-29 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Visuel Analog Scale | From enrollment to the end of treatment at 8 weeks"
  In the evaluation of patient fatigue, patients will be asked to mark on a 100 mm horizontal line. According to VAS, a 0 mm point on this line indicates no fatigue, while a 100 mm point indicates very severe fatigue.
Six Minute Walking Test | From enrollment to the end of treatment at 8 weeks
  It is a test frequently used to evaluate functional capacity. The distance that patients walk in a 30-meter corridor on a flat surface for 6 minutes will be recorded.

SECONDARY OUTCOMES:
PedsQL Multidimensional Fatigue Scale | From enrollment to the end of treatment at 8 weeks
  It is a measurement method consisting of 18 questions developed to evaluate fatigue in pediatric patients.
Fatigue Severity Scale | From enrollment to the end of treatment at 8 weeks
  It is a tool consisting of 9 questions that evaluates fatigue severity.
30 Second Sit-to-Stand Test | From enrollment to the end of treatment at 8 weeks
  One of the tests that will be used to test the functional capacity of individuals is the 30-second sit-to-stand test. During the test, patients will be asked to sit with their hands crossed over their shoulders and their feet touching the ground, and to do a full sit-to-stand in this position. The number of correct standing ups within thirty seconds will be recorded as the test score.
10-Step Climbing Test | From enrollment to the end of treatment at 8 weeks
  In order to evaluate the functional capacity of the patients, they will be asked to quickly climb up and down 10 stairs and the test score will be recorded in seconds.
Half Squat Test | From enrollment to the end of treatment at 8 weeks
  Individuals will be asked to maintain a half squat position on a hard surface, feet shoulder-width apart, hands crossed over shoulders, without shoes, in order to assess their functional capacity. The duration of the squat will be recorded in seconds.
Pacer Run Test | From enrollment to the end of treatment at 8 weeks
  They will be asked to run between two cones in a 20-meter corridor, paying attention to the beeps coming from the voice recorder. The test will start at a slow running speed, and the speed will gradually increase every minute. If individuals cannot reach the cone line the first time when the beep sounds, they will be asked to run in the opposite direction. At the end of the test, the total number of completed laps will be taken as the score, including the laps that were not completed.
Single Leg Stand Test | From enrollment to the end of treatment at 8 weeks
  In order to assess the balance of the subjects, they will be asked to stand on one leg with their hands crossed on their chest and the knee joint flexed at 90 degrees. It will be repeated for both the right and left extremities. The test score will be recorded in seconds.
Functional Forward Reach Test | From enrollment to the end of treatment at 8 weeks
  Individuals will be asked to turn sideways to the wall, flex their arm 90 degrees from the shoulder, and make a fist. The third metacarpophalangeal joint will be marked as the starting point and individuals will be asked to reach forward as much as possible without taking a step or bending their knees. The third metacarpophalangeal joint alignment will be marked again at the last point reached. The distance between the two marked points will be recorded in centimeters.
K- Force-Kinvent Measurement and Evaluation Set | From enrollment to the end of treatment at 8 weeks
  Balance skills will be tested during postures such as squat posture on K-Force plates, single leg and double leg postures with eyes open and closed.
Digitsole Pro Smart Insole System | From enrollment to the end of treatment at 8 weeks
  The walking parameters of individuals will be evaluated with the Digitsole Smart Insole system. Digitsole Pro® smart insole is a valid and reliable measurement tool that allows the individual to evaluate the walking parameters of the individual by being placed inside the shoe worn by the participant. Individuals will be asked to walk wearing smart insoles with sensors inside their shoes. The spatio-temporal and kinematic walking parameters of individuals will be evaluated with the Digitsole Pro system.
FitnessGram Test Battery- Sit-up test | From enrollment to the end of treatment at 8 weeks
  The FitnessGram test battery is a valid and reliable measurement method. Its components include functional capacity, flexibility, muscle strength, body composition and muscular endurance. The FitnessGram test battery will include the Sit-up test, Push-up test, Sit-and-reach test, Trunk lift test and Pacer test. The sit-up test will begin with the patient in a supine position with the knees flexed approximately 140 degrees and the knees slightly apart. The patient will be asked to do sit-ups in accordance with the commands from the voice recorder while the arms are extended next to the body, with the shoulder blades slightly lifted off the ground. The number of sit-ups will be recorded.
FitnessGram Test Battery-The push-up test | From enrollment to the end of treatment at 8 weeks
  The push-up test, individuals will be asked to do push-ups in accordance with the commands from the device with the help of elbow flexion and extension while in the prone position. The number of push-ups done correctly will be recorded. The push-up test provides information about the endurance of the upper extremity muscles.
FitnessGram Test Battery-The Sit-Reach test | From enrollment to the end of treatment at 8 weeks
  The Sit-Reach test: A plate with a length of 50 cm and a width of 45 cm is placed on a box with a length of 35 cm, a width of 45 cm and a height of 32 cm. During the test, individuals will reach forward with their hands as far as they can, with one knee in extension and the other knee in flexion in front of the test box. The evaluation will be repeated for the other side. At the end of the test, the distance the individual reaches will be recorded in cm
FitnessGram Test Battery-The trunk lift test | From enrollment to the end of treatment at 8 weeks
  The trunk lift test will be performed to evaluate trunk extensor muscle endurance. The test will begin with the individual's hands placed under the thighs in a prone position on a flat surface. The subjects will be asked to slowly lift their trunks upwards with their heads. At the end of the test, the distance between the ground and the subjects' chin will be recorded in cm.
FitnessGram Test Battery- body composition | From enrollment to the end of treatment at 8 weeks
  Body mass index will be calculated for body composition.
Visuel Analog Scale | From enrollment to the end of treatment at 8 weeks
  Patients will be asked to mark their pain level on a 100 mm line. 0 mm on the line represents "no pain" and 100 mm represents "very severe pain."

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No